CLINICAL TRIAL: NCT00747669
Title: A Pharmacokinetic Study of Synera™ (Lidocaine 70 mg and Tetracaine 70 mg Topical Patch) to Evaluate the Systemic Exposure to Lidocaine and Tetracaine in Neonates and Infants
Brief Title: Pharmacokinetic Study of Synera™ in Neonates and Infants
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty with enrollment
Sponsor: ZARS Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EN3274-401
Record Dates: First submitted 2008-09-03; First posted 2008-09-05 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Lidocaine; Tetracaine; Transdermal Patch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: lidocaine 70mg and tetracaine 70mg topical patch — One Synera Patch applied for 30 minutes.
  Other Names: Synera

SUMMARY:
This study will measure the amount of lidocaine and tetracaine in the blood after a 30 minute application of Synera.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be an infant of 1 to 4 months of age and weigh at least 2.5 kg or a neonate of 0 to 4 weeks postnatal age with a gestation period of at least 37 weeks, and weigh at least 1.8 kg.
* Subject is scheduled to have a medically indicated minor superficial procedure for which topical local anesthesia would provide a benefit.
* Subject has or will have an indwelling vascular access catheter for blood sampling at the time of the procedure visit. The indwelling vascular access catheter placement must be necessary for medical reasons other than the purposes of this study.
* The additional blood draws for the purposes of this study do not pose more than a minor risk to the health and welfare of the subject.

Exclusion Criteria:

* Subject has known allergies or sensitivities to any component of Synera.
* Subject has clinically significant laboratory abnormalities.
* Subject has known multiple allergies that could indicate hypersensitive skin.
* Subject has known active atopic dermatitis at or near the patch application site.

Max Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Estimated)
Dates: Start 2008-09; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Evaluate the systemic exposure to lidocaine and tetracaine following application of Synera | 30 hours

SECONDARY OUTCOMES:
Monitor the nature and frequency of adverse events | 30 Hours

CONTACTS AND LOCATIONS:
Overall Officials: ZARS Clinical Development, Study Chair — ZARS Pharma
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States